CLINICAL TRIAL: NCT02192931
Title: A Randomized Double-Blind Controlled Trial of Creatine in Female Methamphetamine Users
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Perry Renshaw (Other)
Responsible Party: Sponsor-Investigator, Perry Renshaw, Professor of Psychiatry, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 73034
Record Dates: First submitted 2014-07-15; First posted 2014-07-17 (Estimated); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Depression; Dual Diagnosis; Drug Addiction
MeSH Terms: conditions — Depression; Substance-Related Disorders | interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Creatine monohydrate (Active Comparator): 5 grams of daily creatine monohydrate for 8 weeks
  Interventions: Drug: Creatine monohydrate
- Placebo (Placebo Comparator): 5 g of placebo for 8 weeks
  Interventions: Drug: Creatine monohydrate
- Healthy Control (No Intervention)

INTERVENTIONS:
Drug: Creatine monohydrate
  Arms: Creatine monohydrate; Placebo

SUMMARY:
Methamphetamine (MA) addiction is a public health concern that causes substantial harm to individual users, and imposes an economic burden in the U.S. totaling up to $48.3 billion annually. This study proposes to address a critical aspect of this problem: the lack of any proven, FDA-approved pharmacological treatments for MA users. The proposal combines an intervention designed to improve energy metabolism in the brain, and a neuroimaging technique capable of measuring the neurochemicals that represent cerebral bioenergetic function. The study will replicate and extend a key neuroimaging finding from the investigators recent MA studies: that MA users have decreased phosphocreatine (PCr) levels in the brain, compared to healthy volunteers. Phosphocreatine is the substrate reservoir for the creatine kinase reaction, which reversibly converts PCr into adenosine triphosphate (ATP), the brain's major energy supply, and creatine. Neuronal energy demands are met through a shift in reaction equilibrium, which is designed to maintain the concentration of ATP constant. Research results from the investigators recent study also showed that female MA users have lower brain PCr levels compared to male users. These findings join the converging lines of evidence that MA use is associated with mitochondrial dysfunction, i.e. deficient energy metabolism, in the brain. Frequently, MA users also experience depression, as well as cognitive deficits. Interestingly, both of these entities are also linked to mitochondrial dysfunction in the brain.

The long-term goal of this research program is to define the alterations in brain chemistry that underlie MA use disorders, and to utilize translational magnetic resonance spectroscopy (MRS) neuroimaging to identify rational brain-based treatment targets. Once a hypothesis-driven intervention is identified, MRS can then be further employed in treatment studies, to verify that "target engagement" is achieved. The specific aims of this proposal are an example of this stepwise scientific process: the nutritional supplement creatine will be tested in a randomized, placebo-controlled study of women with MA use disorders, to investigate creatine's effect on cerebral PCr levels, depressive symptoms, and MA usage.

ELIGIBILITY:
Inclusion Criteria:

* Female gender, ages 18-55 inclusive
* Current primary diagnosis of MA dependence or abuse, with MA preferred drug of abuse
* Current diagnosis of Major Depressive Disorder
* Current HAMD score > 15
* Clinical Global Impressions Severity depression score > 4
* If currently taking a psychotropic medication for depressed mood, regimen must be stable for > 4 weeks before randomization

Exclusion Criteria:

* Persons unable to provide adequate consent
* Persons who are at clinically significant suicidal or homicidal risk
* Primary substance-related diagnosis other than MA dependence or abuse
* Comorbid substance dependence diagnosis, other than nicotine (substance abuse diagnoses are not excluded)
* Positive pregnancy test
* Positive test for the antibody to the Human Immunodeficiency Virus (HIV)
* History of renal disease

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2014-09; Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Perry Renshaw, MD, PhD, MBA, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We complied with safety measures meant to minimize the risk of exposure to COVID-19. Participant recruitment were facilitated by advertisements in newspapers, on the radio, by hanging recruitment materials, on the Internet, and by sending letters to social workers and staff at treatment centers. To increase the study's enrollment of healthy controls, we distributed materials specifically aimed at healthy controls.
Groups:
- Creatine Monohydrate: 5 grams of daily creatine monohydrate for 8 weeks
  Creatine monohydrate
- Placebo: 5 g of placebo for 8 weeks
  Creatine monohydrate
- Healthy Control: Measured at baseline.
Period: Overall Study
Arm/Group | Creatine Monohydrate | Placebo | Healthy Control
Started | 21 | 20 | 24
Completed | 12 | 9 | 24
Not Completed | 9 | 11 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Creatine Monohydrate | Placebo | Healthy Control | Total
Number analyzed (Participants) | 21 | 20 | 24 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 20 | 24 | 65
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (7.1) | 34.2 (10.0) | 30.8 (10.5) | 33.8 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 24 | 65
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 18 | 17 | 18 | 53
  Race: Asian | 0 | 0 | 2 | 2
  Race: More than one race | 0 | 0 | 0 | 0
  Race: Native American | 0 | 1 | 0 | 1
  Race: Hispanic/Latino | 3 | 2 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 24 | 65

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale (HAMD) Scores
Description: Change in Hamilton Depression Rating Scale (HAMD) scores will be evaluated over the course of the 8-week treatment period. The HAMD provides an indication of depression and over time provides a valuable guide to progress. Total score ranges from 0 to 54. 0 means no depression and 24 and above means severe depression.
Time Frame: 8-weeks
Population: Due to participant attrition, data analyzed in one or more rows differed from the overall number analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Healthy Control: Healthy Control subjects did not receive study medication.
Arm/Group | Creatine Monohydrate | Placebo | Healthy Control
Number analyzed (Participants) | 20 | 19 | 24
score on a scale
  Screening | 16.76 (3.33) | 17.65 (4.66) | 1.67 (1.90)
  Baseline Scan | 16.24 (3.91) | 14.90 (4.10) | 1.58 (2.21)
  Week 8 Final Scan: number analyzed (Participants) | 12 | 11 | 24
  Week 8 Final Scan | 9.33 (3.58) | 8.18 (7.26) | 1.88 (2.58)

2. Secondary Outcome: Beck Anxiety Inventory (BAI) Scores
Description: Change in Beck Anxiety Inventory (BAI) scores will be evaluated over the course of the 8-week treatment period. The BAI aims to assess the severity of anxiety symptoms, helping clinicians and researchers understand the level of anxiety an individual is experiencing. 0 means minimal anxiety and 30-63 means severe anxiety. The scale ranges from 0 to 63. Total score is reported.
Time Frame: 8-weeks
Population: Due to participant attrition, data analyzed on one or more rows differ from the overall number analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Healthy Control: Health Control subjects did not receive study medication.
Arm/Group | Creatine Monohydrate | Placebo | Healthy Control
Number analyzed (Participants) | 20 | 19 | 24
score on a scale
  Screening | 22.76 (12.70) | 29.25 (12.08) | 3.63 (4.67)
  Baseline | 20.81 (12.00) | 24.60 (13.56) | 4.13 (4.67)
  Week 8 Final Scan: number analyzed (Participants) | 12 | 19 | 24
  Week 8 Final Scan | 6.00 (5.20) | 12.82 (18) | 3.64 (4.23)

3. Other Pre Specified Outcome: BL Neurochemistry Measured by Magnetic Resonance Spectroscopy
Description: Neurochemistry, such as phosphocreatine (PCr), will be measured pre- and post-creatine/placebo treatment.
Time Frame: Baseline
Population: Phosphocreatine (Baseline comparison between creatine and placebo)
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Creatine Monohydrate | Placebo | Healthy Control
Number analyzed (Participants) | 21 | 20 | 0
ratio | 0.268 [0.251 to 0.285] | 0.268 [0.246 to 0.290] |

4. Other Pre Specified Outcome: Neurochemistry Measured by Magnetic Resonance Spectroscopy TX
Description: Neurochemistry, such as phosphocreatine (PCr), will be measured pre- and post-creatine/placebo treatment.
Time Frame: 8-weeks
Population: Phosphocreatine (Treatment comparison between creatine and placebo)
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Creatine Monohydrate | Placebo | Healthy Control
Number analyzed (Participants) | 12 | 9 | 0
ratio | 0.291 [0.265 to 0.317] | 0.269 [0.251 to 0.287] |

ADVERSE EVENTS:
Time Frame: week 8
Description: Participant report
Arm/Group | Creatine Monohydrate | Placebo | Healthy Control
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20 | 0/24
Other Adverse Events (participants affected / at risk) | 3/21 | 7/20 | 0/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Creatine Monohydrate (N=21) | Placebo (N=20) | Healthy Control (N=24)
Diarrhea (Gastrointestinal disorders) | 3 | 7 | 0 — Diarrhea, "Feeling Warm"

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT02192931/Prot_SAP_000.pdf